CLINICAL TRIAL: NCT03572673
Title: Randomized Controlled Multicenter Study to Evaluate the Performance of a New 2-piece Ostomy Appliance vs. Flexima® 3S in Patients With Enterostomy
Brief Title: Study to Evaluate the Performance of a New 2-piece Ostomy Appliance vs. Flexima® 3S in Patients With Enterostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BBraun Medical SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OPM-G-H-1705
Record Dates: First submitted 2018-04-23; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Enterostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexima 3S (Active Comparator): Flexima 3S is a 2-piece ostomy appliance composed with an adhesive base plate and a drainable pouch for collecting stools (1 base plate for 5 days and 1 pouch for 5 days)
  Interventions: Device: Flexima 3S
- New 2-piece ostomy appliance (Experimental): New 2-piece appliance is a 2-piece ostomy appliance composed with an adhesive base plate and a drainable pouch for collecting stools (1 base plate for 5 days and 1 pouch for 5 days)
  Interventions: Device: New 2-piece ostomy appliance

INTERVENTIONS:
Device: Flexima 3S — Flexima 3S (2-piece appliance) with drainable pouch
  Other Names: Class 1 appliance for patients having an enterostoma
  Arms: Flexima 3S
Device: New 2-piece ostomy appliance — New 2-piece ostomy appliance with drainable pouch
  Other Names: Class 1 appliance for patients having an enterostoma
  Arms: New 2-piece ostomy appliance

SUMMARY:
To compare the performance of the comparator Flexima 3S appliance to a new 2-piece appliance in patients with enterostomy.

ELIGIBILITY:
Inclusion Criteria:

* patient having a colostomy or an ileostomy for at least 1 month
* patient currently using a flat appliance
* patient wearing his appliance, on average, at least 5 days
* patient with a stoma's diameter less than 65 mm
* patient who agrees to participate in the evaluation and who have signed the inform consent
* patient having a mental capacity to participate to the study (i.e. to understand the study and to answer to the questions)

Exclusion Criteria:

* Patient currently suffering from peristomal skin complications (bleeding or red and broken skin at the time of inclusion)
* Patient receiving or having received, within the last month, chemotherapy or corticotherapy
* Patient already participating in another clinical study or who have previously participated in this investigation
* Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in base plate wear time, on average every 5 days, up to 21 (±3) days, for each study period | On average every 5 days, up to 21 (±3) days for each period
  For each base plate, the wear time will be evaluated during 21 (±3) days

SECONDARY OUTCOMES:
Assessment of the condition of peristomal skin | After base plate removal at protocol visit 1 (day 0) and visit 2 (at 21 (±3) days)
  Using a standardized measuring ostomy skin tool
Assessment of the main reason of base plate removal | From date of randomization, on average every 5 days, after each base plate removal, up to 21 (±3) days for each study period
  After each base plate removal, the patient will describe on a 7-point scale the main reason of base plate removal ("habit", "hygiene", "leakage under the base plate", "unsticking of the base plate periphery", "unsticking of the base plate, not only on the periphery", "ask for the study but the base plate could stay longer in place", "other, to specify". No value is considered as the better outcome, it's only descriptive value.
Assessment of acceptability | At the end of each study period (21 (±3) days), at visit 2 (21 (±3) days) and at visit 3 (42 (±6) days)
  At the end of each study period (21 (±3) days), the patient will assess on a 4-point scale each parameter of acceptability ("very good", "good", "bad", "very bad". The "very good" value is considered as the better outcome.
Assessment of use of accessories | From date of randomization, on average every 5 days, after each base plate removal, up to 21 (±3) days for each study period
  After each base plate removal, the patient will describe on a 8-point scale the use of accessories ("none", "protective spray", "powder", "paste", "ring", "adhesive remover", "belt", "other, to specify". No value is considered as the better outcome, it's only descriptive value.
Preference between Flexima® 3S and the new 2-piece ostomy appliance | At the end of the study, at 42 (±6) days
  At the end of the study, the patient will notify the preference between Flexima® 3S and the new 2-piece appliance
Safety: Adverse(s) Event(s) | From date of randomization until the date of first adverse event, assessed up to 42 (±6) days
  Description of all adverse event related or not to the devices studied

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Hospital Selayang, Batu Caves
  - Hospital Canselor Tuanku Muhriz, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No